CLINICAL TRIAL: NCT03128164
Title: A Phase 1 Open-Label Study to Assess the Safety, Pharmacokinetics and Preliminary Efficacy of HMPL-689 in Patients With Lymphomas Failed of Standard of Care or No Standard of Care Existed
Brief Title: A Study of HMPL-689 in Patients With Lymphomas Failed of Standard of Care or no Standard of Care Existed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-689-GLOB1
Record Dates: First submitted 2017-03-30; First posted 2017-04-25 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: This study consists of a dose escalation stage (Stage I) and a dose expansion stage (Stage II). Dose escalation will be performed according to a modified toxicity probability interval scheme-2 (mTPI-2). Expansion stage of the study enrolled 143 patients with B cell lymphoma, including CLL/SLL, FL, MZL, DLBCL, MCL and PTCL, Patients were treated with RP2D as starting dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Six arm including in dose expansion stage by following: (Experimental): * Arm A: patients with MZL (subtype including nodal, extra-nodal and splenic) who received ≥ 1 previous line of systematic treatment and at least one line included CD20-directed regimen
  * Arm B: patients with CLL/SLL who received ≥ 1 previous line of systematic treatment and at least one of which included purine-based regimen or CD20-directed regimen
  * Arm C: patients with FL (grade 1, 2, and 3a) who received ≥ 2 previous line of systematic treatment and at least one line included CD20-directed regimen
  * Arm D: patients with MCL who received ≥ 2 previous line of systematic treatment and at least one line included CD20-directed regimen
  * Arm E: patients with DLBCL (including GCB and non-GCB, Richter' transformation) who received ≥ 2 previous line of systematic treatment and at least one line included CD20-directed regimen
  * Arm F: patients with PTCL who received ≥ 2 previous line of systematic treatment
  Interventions: Drug: HMPL-689

INTERVENTIONS:
Drug: HMPL-689 — Two strengths of HMPL-689 capsules (2.5 mg and 10 mg) will be used for clinical studies. The drug products are capsules.

SUMMARY:
This is a Phase 1, open-label study of HMPL-689 administered orally to patients with lymphoma for whom failed of standard care or have no standard of care.This study consists of a dose escalation stage (Stage I) and a dose expansion stage (Stage II).

DETAILED DESCRIPTION:
Both Stage I and Stage II include the following periods: screening period, treatment period, safety follow-up period, and extended progression free survival (PFS) follow-up period, as defined in Dose Escalation Stage (Stage I).

Dose escalation will be performed according to a modified toxicity probability interval scheme-2 (mTPI-2).To further characterize safety and efficacy of HMPL-689 at RP2D, expansion stage of the study enrolled 144 patients with B cell lymphoma, including CLL/ SLL, FL, MZL, DLBCL, MCL and PTCL. Patients were treated with RP2D as starting dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Ability to comply with the protocol
3. Age ≥ 18 years old
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Histologically confirmed lymphoma
6. Relapsed or refractory disease after failed of standard of care or no standard of care existed according to local guideline, and need further systematic treatment in the opinion of the investigator
7. At least 1 bi-dimensionally measurable nodal disease, defined as >1.5 cm (extra-nodal lesion>1.0 cm ) in its largest dimension by computerized tomography (CT) scan is required for patients with lymphoma other than CLL; lesions in anatomical locations (such as extremities or soft tissue lesions) that are not well visualized by CT may be measured by magnetic resonance image (MRI) instead
8. Expected survival of more than 24 weeks
9. Female patients of child-bearing potential and male patients with partners of child-bearing potential must agree to use double barrier contraception, condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD), contraceptives (oral or parenteral), Implanon®, injectable or other avoidance of pregnancy measures during the study and for 30 days after the last day of treatment. Post-menopausal females (>45 years old and without menses for >1 year) and surgically sterilized females are exempt from this criterion

Exclusion Criteria:

1. Patients with CNS(Central nervous system) involvement
2. Any of the following laboratory abnormalities:

   Absolute neutrophil count < 1.5×109/L Hemoglobin <90 g/L Platelets< 100 ×109/L
3. Inadequate organ function, defined by the following:

   Total bilirubin >1.5 x the upper limit of normal (ULN) with the following exception:
   * Patients with known Gilbert's disease who have serum total and direct bilirubin level ≤ 2.5 x the ULN and normal aspartate transaminase (AST) and alanine transaminase (ALT) may be enrolled

   AST or ALT >2.5 x the ULN with the following exception:
   * In the dose expansion stage:Patients with documented disease infiltration of the liver may have AST and ALT levels ≤ 5 x the ULN

   Serum creatinine >1.5 x the ULN or estimated creatinine clearance (Ccr) (i.e., estimated Glomerular Filtration Rate, [eGFR[ according to the method of Cockcroft-Gault )< 60 mL/min
4. International normalized ratio (INR) >1.5 x the ULN or activated partial thromboplastin time (aPTT) >1.5 x the ULN or Prothrombin Time (PT) >1.5 x the ULN
5. Serum amylase or lipase >ULN at screening
6. Patients with presence of second primary malignant tumors within the last 5 years, with the exception of the following non-invasive malignancies after curative treatment:

   Basal cell carcinoma of the skin Squamous cell carcinoma of the skin Carcinoma in situ of the cervix Carcinoma in situ of the breast Asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for≥ 1 year prior to randomization
7. Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, or current known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
8. Prior treatment with any PI3K inhibitors and discontinued due to disease progression
9. Any anti-cancer therapy, including chemotherapy, radiotherapy within 3 weeks prior to initiation of study treatment
10. G-CSF/blood transfusion is prohibited 7 days before the screening hematology test
11. Any steroid therapy or approved targeted small molecule agents for anti-neoplastic intent within 7 days or approximately 5 half-lives, whichever is the longer, prior to initiation of study treatment
12. Any monoclonal antibody for anti-neoplastic intent within 6 weeks or 2 half-lives, whichever is the longer, prior to initiation of study treatment
13. Prior use of any anti-cancer vaccine
14. Prior administration of radioimmunotherapy within 3 months prior to initiation of study treatment
15. Prior use of any drug that is a strong inducer of CYP3A4, strong inhibitor of CYP3A4 within 2 weeks prior to initiation of study treatment (refer to Appendix 13)
16. Prior autologous transplant within 6 months prior to initiation of study treatment
17. Prior allogeneic stem cell transplant within 6 months prior to initiation of study treatment or with any evidence of active graft versus host disease or requirement for immunosuppressants within 21 days prior to initiation of study treatment
18. Clinically significant active infection (e.g., pneumonia)
19. Major surgical procedure within 4 weeks prior to initiation of study treatment
20. Treatment within a clinical study of an investigational agent or using an investigational device within 30 days prior to initiation of study treatment
21. Adverse events from prior anti-cancer therapy that have not resolved to Grade 1, except for alopecia
22. Pregnant (positive pregnancy test) or lactating women
23. New York Heart Association (NYHA) Class II or greater congestive heart failure
24. Congenital long QT syndrome or QTc > 450 msec
25. Currently use medication known to cause QT prolongation or torsades de pointes
26. History of myocardial infarction or unstable angina within 6 months prior to initiation of study treatment
27. History of stroke or transient ischemic attack within 6 months prior to initiation of study treatment
28. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
29. History of inflammatory bowel disease (e.g., Crohn disease or ulcerative colitis)
30. History of drug-induced pneumonitis
31. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Dose limited toxicities evaluated with NCI CTCAE v4.03 | within 28 days after the first dose
  Incidence of dose limited toxicities and associated dose of HMPL-689
Objective response rate (ORR) | Through study completion, 1 year after the last patient has enrolled in the study or all patients have discontinued the study, whichever comes sooner
  Overall response rate (ORR) is defined as the proportion of patients who have a CR or PR

SECONDARY OUTCOMES:
Maximum plasma concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug
Time to reach maximum concentration calculated with Blood samples | within 29 days after the first dose
  Blood samples will be taken to measure the levels of study drug

OTHER OUTCOMES:
Adverse events evaluated by NCI CTCAE v4.03 | from the first dose to within 30 days after the last dose
  Incidence of adverse events and associated dose of HMPL-689
Complete response rate (CR rate) | Through study completion, 1 year after the last patient has enrolled in the study or all patients have discontinued the study, whichever comes sooner
  Complete response rate (CR rate) is defined as the proportion of patients who have a CR Other lymphomas: Lugano Response Criteria for Hodgkin and Non-Hodgkin's Lymphoma [the Revised Response Criteria for Malignant Lymphoma (Cheson 2014)
Time to response (TTR) | Through study completion, 1 year after the last patient has enrolled in the study or all patients have discontinued the study, whichever comes sooner
  Time to response (TTR) is defined as the date from the first dose of study drug to the date of first CR or PR
Duration of response (DoR) | Through study completion, 1 year after the last patient has enrolled in the study or all patients have discontinued the study, whichever comes sooner
  Duration of response (DoR): defined as the time from when the first CR or PR was achieved until the earlier of the first documentation of definitive disease progression or death from any cause Other lymphomas: Lugano Response Criteria for Hodgkin and Non-Hodgkin's Lymphoma [the Revised Response Criteria for Malignant Lymphoma (Cheson 2014)
Clinical benefit rate (CBR): | Through study completion, 1 year after the last patient has enrolled in the study or all patients have discontinued the study, whichever comes sooner
  Clinical benefit rate (CBR): defined as the proportion of patients who have a CR/CRi, PR/PR-L or SD
Progression-free survival (PFS) | Through study completion, 1 year after the last patient has enrolled in the study or all patients have discontinued the study, whichever comes sooner
  Progression-free survival (PFS) is defined as the time from the first dose to the first occurrence of progression or death from any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, MD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - TongJi Medical College Huazhong University of Science& Technology, Wuhan, Hubei
  - Sun Yat-sen University cancer center, Guangzhou
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No